CLINICAL TRIAL: NCT02809196
Title: A Digital Messaging Education Program for Dietary Behavior Modification Towards Healthier Lifestyle Among Danish Adolescents
Brief Title: Texts For Healthy Teens: A Health Education Program for Adolescents
Acronym: T4HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Fetal Programming, Denmark (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Epidemic Health, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2014-01
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Food Habits
Keywords: Food Habits; Adolescents; Digital Communication; BMI
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1: Tailored, friend and mother (Active Comparator): Depending on the responses to the online dietary questionnaire, the tailored SMS-based educational programs can be one out of three different programs, focusing on either sugar sweetened beverages (SSB), fruit and vegetables (F&V), or fish (FISH). About 40 messages will be distributed over 4 weeks.
  Friend and mother are invited to participate.
  Interventions: Behavioral: 1: Tailored SMS program implicating friend and mother
- 2: Standardized, friend and mother (Active Comparator): The standardized SMS-based educational program includes 121 messages there will be distributed over 12 weeks.
  Friend and mother are invited to participate.
  Interventions: Behavioral: 2: Standardized SMS program implicating friend and mother
- 3:Tailored, friend and not mother (Active Comparator): Depending on the responses to the online dietary questionnaire, the tailored SMS-based educational programs can be one out of three different programs, focusing on either sugar sweetened beverages (SSB), fruit and vegetables (F&V), or fish (FISH). About 40 messages will be distributed over 4 weeks.
  Friend is invited to participate but not mother.
  Interventions: Behavioral: 3: Tailored SMS program implicating friend, not mother
- 4: Standardized, friend and not mother (Active Comparator): The standardized SMS-based educational program includes 121 messages there will be distributed over 12 weeks.
  Friend is invited to participate but not mother.
  Interventions: Behavioral: 4: Standardized SMS program implicating friend, not mother
- 5:Tailored, mother and not friend (Active Comparator): Depending on the responses to the online dietary questionnaire, the tailored SMS-based educational programs can be one out of three different programs, focusing on either sugar sweetened beverages (SSB), fruit and vegetables (F&V), or fish (FISH). About 40 messages will be distributed over 4 weeks.
  Mother is invited to participate but not friend.
  Interventions: Behavioral: 5: Tailored SMS program implicating mother, not friend
- 6: Standardized, mother and not friend (Active Comparator): The standardized SMS-based educational program includes 121 messages there will be distributed over 12 weeks.
  Mother is invited to participate but not friend.
  Interventions: Behavioral: 6: Standardized SMS program implicating mother, not friend
- 7:Tailored, not friend, not mother (Active Comparator): Depending on the responses to the online dietary questionnaire, the tailored SMS-based educational programs can be one out of three different programs, focusing on either sugar sweetened beverages (SSB), fruit and vegetables (F&V), or fish (FISH). About 40 messages will be distributed over 4 weeks.
  Neither friend nor mother is invited to participate.
  Interventions: Behavioral: 7: Tailored SMS program not implicating mother or friend
- 8: Standardized, not friend, not mother (Active Comparator): The standardized SMS-based educational program includes 121 messages there will be distributed over 12 weeks.
  Neither friend nor mother is invited to participate.
  Interventions: Behavioral: 8: Standardized SMS program not implicating mother or friend
- 9: No SMS program (Other): Control Group; no SMS-based educational program
  Interventions: Behavioral: 9: No SMS program

INTERVENTIONS:
Behavioral: 1: Tailored SMS program implicating friend and mother
  Arms: 1: Tailored, friend and mother
Behavioral: 2: Standardized SMS program implicating friend and mother
  Arms: 2: Standardized, friend and mother
Behavioral: 3: Tailored SMS program implicating friend, not mother
  Arms: 3:Tailored, friend and not mother
Behavioral: 4: Standardized SMS program implicating friend, not mother
  Arms: 4: Standardized, friend and not mother
Behavioral: 5: Tailored SMS program implicating mother, not friend
  Arms: 5:Tailored, mother and not friend
Behavioral: 6: Standardized SMS program implicating mother, not friend
  Arms: 6: Standardized, mother and not friend
Behavioral: 7: Tailored SMS program not implicating mother or friend
  Arms: 7:Tailored, not friend, not mother
Behavioral: 8: Standardized SMS program not implicating mother or friend
  Arms: 8: Standardized, not friend, not mother
Behavioral: 9: No SMS program
  Arms: 9: No SMS program

SUMMARY:
The overall objective is to examine if participating in an SMS-transmitted health educational program targeting a cluster of dietary factors over a period of weeks during the years of adolescence can induce durable changes towards more healthful dietary habits and body weight trajectories. The investigators will examine if impact is reinforced by asking a friend of the participant to also participate; if impact is reinforced by asking the mother of the participant to also participate; and if impact is reinforced when the SMS-transmitted health promotion program is designed to target a specific dietary factor only - decided upon from participants' reporting of their dietary habits at the beginning of the program - rather than to simultaneously target a cluster of dietary issues uniform for all participants.

DETAILED DESCRIPTION:
Groups of adolescents from the Danish National Birth Cohort (DNBC) will be offered to participate in the health educational programs. At 14 years and 14 years plus 3 months all children DNBC are invited to report comprehensively on their dietary and physical activity habits by means of a web-based questionnaire (FFQ). Eligible DNBC adolescents for the SMS-educational program will be invited among those who have completed the FFQ. Thus, once they have completed the DNBC FFQ, they may be invited to participate in the SMS-based educational programs, either addressing only one of the three target factors: sugar sweetened beverages, fruit & vegetables, or fish (SSB, F&V, or Fish) or addressing all three factors (cluster). The adolescents may also potentially be invited to include a friend, their mother or both.

Trial Organization:

* Sjurdur F Olsen, MD PhD, Lead Principal Investigator (Responsible Party), Statens Serum Institut, Copenhagen, Denmark;
* Eric Ding, ScD, Co-PI, Harvard TH Chan School of Public Health;
* Daniel Zoughbie, Co-PI, Epidemic Health Inc.

Design for Inviting Adolescents to Educational Program: The study will be conducted corresponding to a '2x2x2 factorial plus 1' design, with 9 arms. In addition to allowing testing of the effect of participating in an SMS based educational program as compared to not participating in such program, this will allow for additional testing of effect of implicating a friend v. not implicating friend; of implicating the mother v. not implicating the mother; and of delivering tailored messaging targeting only one of the three dietary factors (SSB, F&V, or Fish) v. delivering uniform messaging targeting all three factors.

In the tailored program, the participants will receive messages distributed over 4 weeks, whereas in the FULL program (addressing all three clusters) messages are distributed over 12 weeks. Messages can be divided into five categories: Information, quizzes, tips, challenges, and reminders.

Hypotheses to tested:

1. Overall effect. Hypothesis 1: SMS messaging (versus being allocated the group not offered to participate in an SMS messaging program) will improve dietary habits and body weight trajectories
2. Effect of including a friend. Hypothesis 2: Including a friend (versus not including a friend) will increase above effects
3. Effect of including the mother. Hypothesis 3: Including the mother (versus not including the mother) will increase above effects
4. Effect of tailored program v. a cluster of factors. Hypothesis 4: A tailored program will be more efficient than a full program in changing specific outcome.

For testing the hypothesis 4, which addresses one of the three specific, tailored programs (underlined below), eligible adolescents will be stratified into four strata depending on their FFQ response:

Stratum 1: Nearly all participants have a low intake of fish; whereas there will be no problem with sugar sweetened beverages and no problem with fruit and vegetables. Tailored program AND outcome measure to be tested: FISH / fish intake.

Stratum 2: All participants have problems with fruit and vegetables, and no problems with sugar sweetened beverages, but (NB!), like in stratum 1, nearly all have a problem with fish. Tailored program AND outcome measure to be tested: F&V / intake fruit and vegetable.

Stratum 3: All participants have problems with sugar sweetened beverages; whereas nearly all will have NO problem with fruit and vegetables. Nearly all have a problem with Fish (986/1195). Tailored program AND outcome measure to be tested: SSB / intake of sugar sweetened beverages.

Stratum 4: All participants have a problem with sugar sweetened beverages, fruit and vegetables and fish. Tailored program AND outcome measure to be tested: FISH / fish intake.

Strata 1 & 4 can be aggregated and, when effect on fish intake is tested, a test for interaction by intake of sugar sweetened beverages or by intake of fruit and vegetables can be made.

A detailed a priori Statistical Analysis Plan SAP (version 2.0) was filed at the Office of Research Integrity, Statens Serum Institut, on June 17, 2019. This date preceded the date of opening the data (i.e., relating the outcome measures to information about which trial arms the adolescents had been randomly allocated to).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents participating in the Danish National Birth Cohort

Exclusion Criteria:

* Lacking information from maternal interviews 1 and 2

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7890 (Actual)
Dates: Primary Completion 2018-10-06 (Actual); Study Completion 2018-10-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in an index reflecting overall dietary quality | 6 months and 18 months after allocation
  Based on reported intake in online questionnaires
Change from baseline in BMI z-score | 6 months and 18 months after allocation
  Based on reported height and weight in online questionnaires

SECONDARY OUTCOMES:
Change from baseline in intake of sugar sweetened beverages | 6 months and 18 months after allocation
  Based on reported intake in online questionnaires
Change from baseline in intake of fruits and vegetables | 6 months and 18 months after allocation
  Based on reported intake in online questionnaires
Change from baseline in intake of fish | 6 months and 18 months after allocation
  Based on reported intake in online questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sjurdur F Olsen, Ph.D., Principal Investigator — Statens Serum Institut; Eric Ding, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Daniel Zoughbie, Principal Investigator — Epidemic Health, Inc.
Locations (1):
- Statens Serum Institut, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjerregaard AA, Zoughbie DE, Hansen JV, Granstrom C, Strom M, Halldorsson ThornI, Meder IK, Willett WC, Ding EL, Olsen SF. An SMS chatbot digital educational program to increase healthy eating behaviors in adolescence: A multifactorial randomized controlled trial among 7,890 participants in the Danish National Birth Cohort. PLoS Med. 2024 Jun 14;21(6):e1004383. doi: 10.1371/journal.pmed.1004383. eCollection 2024 Jun. PMID 38875292